CLINICAL TRIAL: NCT03007784
Title: Two Intensities of Transcranial Direct Current Stimulation to Improve Consciousness in Severely Brain Injured Patients
Acronym: STIMCOM
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Groupe Hospitalier Pitie-Salpetriere (Other)
Collaborators: Hôpital Raymond Poincaré (Other); Hospices Civils de Lyon (Other)
Responsible Party: Principal Investigator, LIONEL NACCACHE, MD, PhD, Groupe Hospitalier Pitie-Salpetriere
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SC20160427
Record Dates: First submitted 2016-12-22; First posted 2017-01-02 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Disorder of Consciousness; Minimally Conscious State; Vegetative State; Cognitive Impairment
Keywords: Consciousness; Disorder of consciousness; Minimally conscious state; Vegetative state; Exit-MCS; Transcranial direct current stimulation (tDCS); CRS-R; EEG; Cognitive ERPs
MeSH Terms: conditions — Consciousness Disorders; Persistent Vegetative State; Cognitive Dysfunction | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 mA anodal tDCS stimulation (Experimental): Anodal tDCS stimulation at 2 mA applied to the left dorsolateral prefrontal during 20 minutes five days a week for two consecutive weeks
  Interventions: Device: transcranial direct current stimulation (tDCS) / Comparison of current intensities
- 0.2 mA anodal tDCS stimulation (Active Comparator): Anodal tDCS stimulation at 0.2 mA applied to the left dorsolateral prefrontal during 20 minutes five days a week for two consecutive weeks
  Interventions: Device: transcranial direct current stimulation (tDCS) / Comparison of current intensities

INTERVENTIONS:
Device: transcranial direct current stimulation (tDCS) / Comparison of current intensities

SUMMARY:
Limited treatments are available to improve consciousness in severely brain injured patients. Transcranial Direct Current stimulation (tDCS) is one of the few therapeutics that showed evidence of efficacy to increase level of consciousness and functional communication in some minimally conscious state (MCS) patients, and in some vegetative state (VS) patients. However the optimal intensity of electrical current stimulation remains unknown.

This study will test the effects of two intensities of tDCS stimulation (either 0.2mA or 2mA) applied on left dorso-lateral prefrontal cortex on both behavior, - assessed by the Coma Recovery Scale-Revised (CRS-R) scores -, as well as quantified EEG recorded during resting state (using algorithms previously designed and published by the investigators) and event-related potentials (using auditory paradigms we previously published) in severely brain damaged patients with disorders of consciousness (MCS, VS, and conscious but cognitively disabled patients) of various etiologies.

DETAILED DESCRIPTION:
This study will use a cross-over double-blind design with each patient receiving both current intensities in a randomized order during 4 weeks (2 weeks for each tDCS intensity, totalizing a number of 10X2 stimulation sessions of 20 minutes each).

ELIGIBILITY:
Inclusion Criteria:

* Non communicative patients (including conscious patients but presenting with major fluctuations of vigilance and/or of cognitive abilities)
* Patients with stable clinical examination
* Age between 18 and 80 years
* Brain injury confirmed by cerebral imaging (MRI or TDM)
* Disorder of consciousness diagnosed by CRS-R (VS, MCS, exitMCS)

Exclusion Criteria:

* Status epilepticus
* Severely neurodegenerative illnesses (Alzheimer disease, Lewy Body Dementia)
* Pregnancy
* Patients underage

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2017-01; Primary Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Change of the Coma Recovery Scale-Revised score according to tDCS current intensity (2mA versus 0.2mA) | Last Day of 0.2mA session (Day 14th or Day 28th) versus Last Day of 2mA session (Day 14th or Day 28th)
  Comparison of the CRS-R score at the tenth day of 0.2mA stimulation (Day14 or Day28) with the score at the tenth day of 2mA stimulation (Day14 or Day28)
Change from baseline of the Coma Recovery Scale-Revised score after 2mA tDCS current intensity | Last Day of 2mA session (Day 14th or Day 28th) versus baseline (Day 1st)
  Comparison of the CRS-R score at the tenth day of 2mA stimulation (Day14 or Day28) with the score at baselne (Day1)
Change from baseline of the Coma Recovery Scale-Revised score after 0.2mA tDCS current intensity | Last Day of 0.2mA session (Day 14th or Day 28th) versus baseline (Day 1st)
  Comparison of the CRS-R score at the tenth day of 0.2mA stimulation (Day14 or Day28) with the score at baselne (Day1)

SECONDARY OUTCOMES:
IChange of the ERPS recorded during the "local global" auditory paradigm (Bekinschtein et al., PNAS 2009) after 10 days of 2mA tDCS current intensity and after 10 days of 0.2mA tDCS current intensity | Last Day of 2mA session (Day 14th or Day 28th) versus Last Day of 0.2mA session (Day 14th or Day 28th)
  Statistical comparison of local (MMN, automatic CNV) and global (P3b; modulation of CNV) ERP effects recorded after 10 days of 2mA tDCS stimulation (Day 14th or Day 28th) and after 10 days of 0.2mA tDCS stimulation (Day 14th or Day 28th)
Change from baseline of the ERPS recorded during the "local global" auditory paradigm (Bekinschtein et al., PNAS 2009) after 2mA tDCS current intensity | Last Day of 2mA session (Day 14th or Day 28th) versus baseline (Day 1st)
  Statistical comparison of local (MMN, automatic CNV) and global (P3b; modulation of CNV) ERP effects recorded at baseline (Day 1) and after 10 days of 2mA tDCS stimulation
Change from baseline of the ERPS recorded during the "local global" auditory paradigm (Bekinschtein et al., PNAS 2009) after 0.2mA tDCS current intensity | Last Day of 0.2mA session (Day 14th or Day 28th) versus baseline (Day 1st)
  Statistical comparison of local (MMN, automatic CNV) and global (P3b; modulation of CNV) ERP effects recorded at baseline (Day 1) and after 10 days of 0.2mA tDCS stimulation
IChange of the multivariate automatic classification of conscious state from EEG (Sitt et al., Brain et al. 2014) after 10 days of 2mA tDCS current intensity and after 10 days of 0.2mA tDCS current intensity | Last Day of 2mA session (Day 14th or Day 28th) versus Last Day of 0.2mA session (Day 14th or Day 28th)
  Statistical comparison of the multivariate automatic classification of conscious state from EEG (Sitt et al., Brain 2014) after 10 days of 2mA tDCS stimulation (Day 14th or Day 28th) and after 10 days of 0.2mA tDCS stimulation (Day 14th or Day 28th)
Change from baseline of the multivariate automatic classification of conscious state from EEG (Sitt et al., Brain et al. 2014) after 10 days of 2mA tDCS current intensity | Last Day of 2mA session (Day 14th or Day 28th) versus baseline (Day 1st)
  Statistical comparison of the multivariate automatic classification of conscious state from EEG (Sitt et al., Brain 2014) at baseline (Day 1st) and after 10 days of 2mA tDCS stimulation (Day 14th or Day 28th) and after 10 days of 2mA tDCS stimulation (Day 14th or Day 28th)
Change from baseline of the multivariate automatic classification of conscious state from EEG (Sitt et al., Brain et al. 2014) after 10 days of 0.2mA tDCS current intensity | Last Day of 0.2mA session (Day 14th or Day 28th) versus baseline (Day 1st)
  Statistical comparison of the multivariate automatic classification of conscious state from EEG (Sitt et al., Brain 2014) at baseline (Day 1st) and after 10 days of 2mA tDCS stimulation (Day 14th or Day 28th) and after 10 days of 0.2mA tDCS stimulation (Day 14th or Day 28th)

CONTACTS AND LOCATIONS:
Overall Officials: Lionel Naccache, MD PhD, Study Director — Paris 6 University ICM Inserm APHP
Locations (1):
- Groupe Hospitalier Pitié-Salpêtrière, Paris, France